CLINICAL TRIAL: NCT01462864
Title: StructUred eduCation Programme to Improve Cardiovascular Risk in womEn With polycyStic Ovary Syndrome; SUCCESS Study
Brief Title: Development of a Structured Education Programme for Women With Polycystic Ovary Syndrome
Acronym: SUCCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: Society for Endocrinology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0209
Record Dates: First submitted 2011-10-18; First posted 2011-11-01 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2011-10

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Lifestyle; Structured Education; Walking Activity; Exercise; Overweight; Impaired Glucose Regulation; Diabetes Prevention
MeSH Terms: conditions — Polycystic Ovary Syndrome; Motor Activity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Lifestyle education intervention
  Interventions: Behavioral: Structured Lifestyle Education
- Control (No Intervention): The control group will receive an information leaflet which is generally distributed in our speciality clinic to patients with diagnosis of PCOS. The leaflet includes general information on PCOS, treatment options and advice on increasing physical activity.

INTERVENTIONS:
Behavioral: Structured Lifestyle Education — A 3-4 hours group education delivered in a patient group composed of 4-8 patients and delivered by two healthcare professionals.
  Arms: Intervention

SUMMARY:
Polycystic Ovary syndrome (PCOS) is a common hormonal imbalance affecting about 12% of women in the UK. The number of women with PCOS is rising. They suffer from a combination of symptoms including excess hair, irregular/absent periods, and infertility. About 70% of women with PCOS are obese or overweight, 10% develop type 2 diabetes (T2DM), and 30-40% have some degrees of abnormality in controlling (metabolising) blood sugar. Studies have shown that if women with PCOS make change to their lifestyle (diet and activity), they may reduce their risk of getting diabetes and heart disease in the future. This study aims to develop and test a programme that can be run in groups (structured education), to support women with PCOS make the lifestyle changes needed to improve their PCOS and prevent future associated health problems. Structured education programmes are suitable for use within the NHS and are already recommended for individuals with T2DM, but have not been tested as a method of treatment for PCOS which is a high risk condition for T2DM.

The investigators aim to initially develop a specific education programme for women with PCOS using their expertise in their disease and defining their needs. The next step is to test this programme on 160 women with PCOS who will be selected from the investigators database or clinics. They will be divided randomly to two groups to receive either this programme or routine care.

The investigators will give them an accelerometer (a very small portable device). This will measure their physical activity and counts their daily steps. The investigators aim is to increase their step count by at least 2000 steps per day after one year.

The investigators believe that the group given the structured education will show some evidence of improvement in their glucose metabolism, and consequently decreased chance of developing diabetes.

DETAILED DESCRIPTION:
Overview of project plan:

Development of the structured education course: Year 1 (Phases 1&2)

Phase 1:

The SUCCESS intervention (structured education programme to improve cardiovascular risk in women with PCOS) will be developed and piloted in line with the Medical Research Council's framework for complex interventions. This will involve recruiting participants for focus groups and interviews to allow the research group to develop a detailed understanding of what the requirements of the structured education course are.

Inclusion criteria for patients in this phase is women with a clear diagnosis of PCOS based on Rotterdam 2003 Criteria or National Institute of Health 1992 And 18< age <70 years Participants will be recruited from a database of patients in our speciality clinic and also primary care if needed and the interviews/ focus groups will be held in locations close to the participant, or over the telephone.

Analysis of these sessions will provide invaluable data for the development of the structured education course.

As part of this phase of the study we will perform a systematic review of the literature on the previous lifestyle interventions in the PCOS.

We will also perform a demographic analysis of almost 2400 patients with diagnosis of PCOS in University Hospitals of Leicester database. We already have the ethical approval for the conducting routine database linkage studies including a linkage with the hospital admission database in local Health Informatics Service. Demographic distribution of diagnosis, complications of PCOS, cardiovascular outcomes, and reported comorbidities besides other information such as deprivation score will inform us of the important issues need to be considered in development of an education intervention for women with PCOS in phase 2 and 3.

Phase 2

Once the course has been designed, it will be piloted in one or two groups of women with PCOS to get feedback on the content and delivery. These feedbacks will be incorporated in the course and contents will be refreshed and refined.

For the above mentioned pilot sessions, patients will only attend a 3.5 hours education session and no test or measurement will be done.

After each session their views on the content and delivery of the education will be sought. We will continue to run these pilot sessions until we get no further new comments. Previous experience with other similar interventions has shown that two pilot sessions are enough.

When the education programme is ready we can test its efficacy in a randomised controlled trial.

Phase 3; Randomised controlled trial: Years 2 & 3

The primary hypothesis of the randomised controlled trial is:

"Structured education can increase physical activity measured as walking steps in women with polycystic ovary syndrome."

Study design:

This is a randomised controlled community based trial. Participants will be randomised to either the intervention or control group at the beginning. A controlled design for the current study is essential given that it is unknown whether structured education is effective at initiating a lifestyle change and whether it translates into improvements in important markers of metabolic and vascular health. Therefore in order to inform health policy evidence is needed from high quality randomized controlled trials carried out in a community setting.

Our study intervention will not interfere with the routine care of a woman diagnosed with PCOS, whether the patient is recruited from speciality clinics or in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Females aged between 18-50 years with the diagnosis of PCOS according to Rotterdam Criteria 2003 who are Overweight: (WHO 2010)

  * Body Mass Index ≥ 23 kg/m2 for Black and Minor Ethnicities
  * Body Mass Index ≥ 25 kg/m2 for White Europeans
* If already on medical treatment for their PCOS, they should be on a stable regime for at least 6 months prior to the recruitment.

Exclusion Criteria:

* Physical condition which limits full participation in the study
* Active psychotic illness or a significant illness which, in the view of the investigators, would prevent full participation
* Inability to communicate in verbal and written English
* Steroid use
* Diabetes
* Pregnancy
* Involvement in other research studies with similar nature

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
we aim for a 2000 steps increase in Number of steps per day | One year
  It has been shown that 1 mmol/L drop in 2 hours glucose tolerance test following lifestyle intervention is significantly effective in diabetes prevention equal to 50% reduction in progression to T2DM. A previous similar intervention in people with IGR by our group in Leicester achieved a significant drop of 1.31 mmol/L (SD 2 mmol/L) in 2 hours glucose tolerance through an increase of 2000 steps per day in walking activity (SD 4000 steps/day).

SECONDARY OUTCOMES:
Physical Activity | One year
  Physical activity will be objectively measured using the accelerometer and also IPAQ.
Biochemical variables | One year
  * Oral glucose tolerance test
  * Blood lipid profile, liver and Kidney function test, albumin, vitamin D, calcium and full blood count.
  * Hormonal assay; Follicular Stimulating Hormone (FSH), Luteinizing Hormone (LH), Testosterone, Sex Hormone Binding Globulin (SHBG), Dehydroepiandostrone (DHEAS), and Androstendione. Day 21 Progesterone level (unless on ovulation suppression medication).
  * Insulin, HbA1c, HOMA-B, HOMA-IR
  * hsCRP, TNF alpha, IL-6, and sIL-6R, fibrinogen, adiponectin
Anthropometric and demographic | One year
  * Blood pressure
  * Body weight
  * Body fat percentage
Health Related Quality of Life | One Year
  PCOSQ is the only specified health related quality of life questionnaire developed and tested for this condition (Cronin 1998), which has been validated in UK (Jones 2004). It contains 26 items measuring 5 areas; emotions, body hair, weight, infertility problems, and menstrual problems.
Exercise and Barrier Self Efficacy | One Year
  It will be measured using the 100% confidence rating scale (from 0% = no confidence to 100% = complete confidence) (Keller 1999). This self-efficacy questionnaire measures participants' confidence in their ability to undertake any form of moderate- to vigorous-intensity physical activity for 10 minute periods, increasing incrementally from 10 minutes to one hour each day. An overall score is calculated by summing the efficacy scores for each time period and dividing by the number of time periods.
Epworth Sleepiness Scale | One Year
  The risk of Obstructive Sleep Apnoea (OSA) has been reported to be 5 to even 30 fold higher in women with PCOS (Nitsche 2010). Epworth Sleepiness Scale is the standard questionnaire developed for clinical assessment of behavioural morbidity associated with OSA and can assess the degree of sleepiness reliably as an screening tool. (Doghramii 2008).
Body Fat Composition | One Year
  In a sub-study of the SUCCESS study population, a whole body dual energy X-ray absorptiometry (DEXA) scan and a single section abdominal magnetic resonance imaging (MRI) scan taken in the L3-L4 region will be used to measure soft tissue body composition and visceral and subcutaneous abdominal fat distribution respectively.
Brief Illness Perception | One Year
  This nine item validated instrument uses an 11 point Likert scale (0 = no effect, 10 = complete effect) to measure five cognitive illness representations (consequences, timeline, personal control, treatment control, and identity), two emotional representations (concern and emotion) and illness comprehensibility (perceived knowledge). The BIPQ has been shown to have reasonable test-retest reliability and concurrent validity (Broadbent 2006).

CONTACTS AND LOCATIONS:
Overall Officials: Melanie J Davies, Prof (MD), Principal Investigator — University of Leicester; Kamlesh Khunti, Prof (PhD), Study Chair — University of Leicester; Hamidreza Mani, MD, Study Director — University of Leicester
Locations (1):
- University Hospitals of Licester, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No